CLINICAL TRIAL: NCT01652690
Title: Prospective Observational Study to Describe Characteristics and Management of Patients With Postmenopausal Osteoporosis Treated With Prolia® in Routine Clinical Practice
Brief Title: Prospective Observational Study to Describe Characteristics and Management of Patients Treated With Denosumab (Prolia®) in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: One Amgen Center Drive (Unknown); THOUSAND OAKS (Unknown); CA (Unknown); 91320-1799 (Unknown); USA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20110132
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Denosumab: Patients with postmenopausal osteoporosis (PMO) who received at least 1 injection of denosumab 60 mg subcutaneously in the Czech Republic and Slovakia.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — This is an non-interventional study, therefore denosumab is administered as part of routine care and not for purposes of the study.
  Other Names: Prolia®

SUMMARY:
The objective of this prospective, observational study in Czech Republic and Slovakia is to describe per country the characteristics of women treated with denosumab in routine clinical practice and the clinical management of these patients during the first 2 years of treatment. In addition, the study aims to collect safety data in the real-life clinical practice settings on adverse drug reactions (ADRs) and serious ADRs.

ELIGIBILITY:
Inclusion Criteria

* Women with a clinical diagnosis of postmenopausal osteoporosis
* Decision has been made to treat with denosumab 60 mg once every 6 months
* Have received their first injection of denosumab within 8 weeks prior to enrolling in this study.
* Appropriate written informed consent has been obtained (as required per local country regulations)

Exclusion Criteria

* Participating in ongoing or have participated in previous denosumab clinical trials
* Participation in other clinical or device trials in the last 6 months
* Contra-indicated for treatment with Prolia® according to the approved applicable local product label.
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted at various study centers in the Czech Republic and Slovakia. Postmenopausal women with osteoporosis who receive an injection of denosumab and meet the inclusion/exclusion criteria will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (26):
- Czechia (14):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Havlíčkův Brod
  - Research Site, Karlovy Vary
  - Research Site, Kutná Hora
  - Research Site, Ostrava
  - Research Site, Ostrava-Trebovice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Trutnov
  - Research Site, Vsetín
  - Research Site, Zlín
  - Osteocentrum Zlin, Zlín
- Slovakia (12):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Humenné
  - Research Site, Kosice-Saca
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Trnava
  - Research Site, Žilina

REFERENCES:
- [Background] Ruzickova O, Killinger Z, Kasalicky P, Hamilton L, Tyl R, Tomkova S, Kalouche-Khalil L. Real-world Management of Women with Postmenopausal Osteoporosis Treated with Denosumab: A Prospective Observational Study in the Czech Republic and Slovakia. Adv Ther. 2018 Oct;35(10):1713-1728. doi: 10.1007/s12325-018-0779-9. Epub 2018 Sep 6. PMID 30191465
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at various study centers in the Czech Republic and Slovakia.
  The recruitment period was from 26 June 2012 to 15 May 2013.
Groups:
- Czech Republic: Patients in the Czech Republic with postmenopausal osteoporosis who received at least 1 injection of denosumab 60 mg administered subcutaneously every 6 months as part of their routine clinical care.
- Slovakia: Patients in Slovakia with postmenopausal osteoporosis who received at least 1 injection of denosumab 60 mg administered subcutaneously every 6 months as part of their routine clinical care.
Period: Overall Study
Arm/Group | Czech Republic | Slovakia
Started | 300 | 300
Completed | 265 | 279
Not Completed | 35 | 21
Not completed — Withdrawal by Subject | 16 | 4
Not completed — Other | 8 | 9
Not completed — Lost to Follow-up | 6 | 6
Not completed — Death | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Czech Republic | Slovakia | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.7) | 64.3 (8.6) | 66.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 300 | 600
  Male | 0 | 0 | 0
Age at Menopause [Mean (Standard Deviation); unit: years] | 48.3 (5.6) | 48.3 (5.2) | 48.3 (5.4)
Time Since Postmenopausal Osteoarthritis Diagnosis [Mean (Standard Deviation); unit: years] | 5.3 (5.2) | 3.0 (4.1) | 4.1 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving All Prescriptions and Injections of Denosumab From the Initial Prescribing Physician's Office
Description: Number of participants who received all injection(s), including baseline injection, from the initial prescribing site irrespective of total number of injections received on study.
Time Frame: 24 months
Population: Full analysis set (all enrolled patients who provided informed consent and received at least one injection)
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants | 295 | 296

2. Primary Outcome: Number of Participants Receiving an Individual Prescription and Injection of Denosumab From the Initial Prescribing Physician Office by Each Individual Injection
Time Frame: Baseline (day 1), and at Months 6, 12, 18 and 24 (corresponding to the first, second, third and fourth post-baseline injections respectively)
Population: Full analysis set; n = the number of participants who received the corresponding injection
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  Baseline injection (n = 300, 300) | 300 | 298
  First post-baseline injection (n = 283, 293) | 282 | 291
  Second post-baseline injection (n = 276, 283) | 275 | 282
  Third post-baseline injection (n = 262, 276) | 260 | 274
  Fourth post-baseline injection (n = 246, 243) | 245 | 240

3. Primary Outcome: Number of Participants Receiving All Prescriptions and Injections of Denosumab
Description: Number of participants receiving all prescriptions and injections of denosumab whether or not the injections are given at the initial prescribing physician's office.
Time Frame: Months 6, 12, 18 and 24 (corresponding to the first, second, third and fourth post-baseline injections respectively)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  First post-baseline injection | 283 | 293
  Second post-baseline injection | 276 | 283
  Third post-baseline injection | 262 | 276
  Fourth post-baseline injection | 246 | 243

4. Primary Outcome: Number of Participants With a Referral by the Prescribing Physician to Other Health Care Providers for Continuation or Follow-up of Care
Time Frame: 24 months
Population: Full analysis set participants who discontinued the study prematurely
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 35 | 21
participants
  Referred to other health care providers (total) | 0 | 2
  Referred to rheumatologist | 0 | 2

5. Primary Outcome: Types of Health Care Providers Administering an Individual Injection of Denosumab at the Baseline Injection
Description: Types of health care providers administering an individual injection of denosumab inside or outside the initial prescribing office at the baseline injection.
Time Frame: Baseline (day 1)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  Prescribing Physician | 54 | 84
  Other Physician | 19 | 21
  Nurse | 227 | 195

6. Primary Outcome: Types of Health Care Providers Administering Denosumab at the First Post-baseline Injection
Description: Types of health care providers administering an individual injection of denosumab inside or outside the initial prescribing office at the first post-baseline injection.
Time Frame: Month 6
Population: Full analysis set participants who received a first post-baseline injection (i.e. at month 6)
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 283 | 293
participants
  Prescribing Physician | 70 | 109
  Other Physician | 8 | 0
  Nurse | 205 | 184

7. Primary Outcome: Types of Health Care Providers Administering Denosumab at the Second Post-baseline Injection
Description: Types of health care providers administering an individual injection of denosumab inside or outside the initial prescribing office at the second post-baseline injection.
Time Frame: Month 12
Population: Full analysis set participants who received a second post-baseline injection (i.e. at month 12)
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 276 | 283
participants
  Prescribing Physician | 75 | 104
  Other Physician | 0 | 0
  Nurse | 201 | 179

8. Primary Outcome: Types of Health Care Providers Administering Denosumab at the Third Post-baseline Injection
Description: Types of health care providers administering an individual injection of denosumab inside or outside the initial prescribing office at the third post-baseline injection.
Time Frame: Month 18
Population: Full analysis set participants who received a third post-baseline injection (i.e. at month 18)
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 262 | 276
participants
  Prescribing Physician | 69 | 113
  Other Physician | 4 | 1
  Nurse | 189 | 162

9. Primary Outcome: Types of Health Care Providers Administering Denosumab at the Fourth Post-baseline Injection
Description: Types of health care providers administering an individual injection of denosumab inside or outside the initial prescribing office at the fourth post-baseline injection.
Time Frame: Month 24
Population: Full analysis set participants who received a fourth post-baseline injection (i.e. at month 24)
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 246 | 243
participants
  Prescribing Physician | 76 | 93
  Other Physician | 0 | 6
  Nurse | 170 | 144

10. Primary Outcome: Number of Denosumab Post-baseline Injections Received by Each Participant
Time Frame: 24 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  No post-baseline injections | 17 | 7
  One post-baseline injection | 7 | 10
  Two post-baseline injections | 14 | 7
  Three post-baseline injections | 16 | 33
  Four post-baseline injections | 246 | 243

11. Primary Outcome: Number of Participants Having Radiologic Bone Assessments
Description: Number of participants having radiologic bone assessments pre-treatment with denosumab and during the study.
Time Frame: Pre-baseline (before first denosumab injection) and during the study (post-baseline)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  Pre-baseline | 297 | 299
  Post-baseline | 253 | 216

12. Primary Outcome: Number of Participants Having Osteoporosis Related Laboratory Examinations
Description: Number of participants having osteoporosis related laboratory examinations pre-treatment with denosumab and during the study. Participants may not have been given denosumab injection when they attended each visit.
Time Frame: Pre-baseline (before first denosumab injection) and post-baseline
Population: Full analysis set; n = participants with visits at each time point.
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  Baseline injection (n = 300, 300) | 230 | 260
  First post-baseline injection (n = 285, 294) | 148 | 207
  Second post-baseline injection (n = 280, 286) | 162 | 224
  Third post-baseline injection (n = 270, 280) | 163 | 226
  Fourth post-baseline injection (n = 262, 263) | 174 | 223

13. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs) to Denosumab
Description: Adverse events (AEs) that were considered related to denosumab as evaluated by the investigator were classified as adverse drug reactions (ADRs).
Time Frame: 24 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  All adverse drug reactions | 4 | 12
  ADRs leading to discontinuation of denosumab | 2 | 5
  Fatal adverse drug reactions | 0 | 0

14. Secondary Outcome: Number of Participants With Serious ADRs to Denosumab
Description: Serious adverse events that were considered related to denosumab were classified as serious adverse drug reactions (SADRs). A serious adverse event (SAE) is any AE that also: • is fatal • is life threatening (places the patient at immediate risk of death) • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • is an "other significant medical hazard" that does not meet any of the above criteria.
Time Frame: 24 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Czech Republic | Slovakia
Number analyzed (Participants) | 300 | 300
participants
  All serious adverse drug reactions | 0 | 1
  SADRs leading to discontinuation of denosumab | 0 | 0
  Fatal serious ADRs | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse drug reactions that exceed the indicated frequency threshold.
  Serious Adverse Events summarizes serious adverse drug reactions which are defined as serious adverse events that are considered related to denosumab.
Arm/Group | Czech Republic | Slovakia
Serious Adverse Events (participants affected / at risk) | 0/300 | 1/300
Other Adverse Events (participants affected / at risk) | 0/300 | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Czech Republic (N=300) | Slovakia (N=300)
Myocardial infarction (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.